CLINICAL TRIAL: NCT00397215
Title: Evaluate Immunogenicity & Safety of a Single or Double-dose of the Pandemic Influenza Candidate Vaccine (GSK1562902A) Given Following a Two-administration Schedule (21 Days Apart) in Adults Over 60 Yrs
Brief Title: Evaluate Safety & Immunogenicity of a Pandemic Influenza Vaccine (GSK1562902A) in Adults Over 60 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 108251; 108252 (Other: GSK); 111275 (Other: GSK); 111276 (Other: GSK); 2006-004041-42 (EudraCT Number)
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-02

CONDITIONS: Influenza
Keywords: H5N1; influenza; vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2; fluarix

ARMS (4):
- GSK1562902A 1 Group (Experimental): Subjects aged 61 years or older at the time of first vaccination received 1 dose of GSK1562902A adjuvanted vaccine at Day 0. The vaccine was administered intramuscularly, in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1562902A) (adjuvanted or not); Biological: Fluarix
- GSK1562902A 2 Group (Experimental): Subjects aged 61 years or older at the time of first vaccination received 1 dose of GSK1562902A non-adjuvanted vaccine at Day 0. The vaccine was administered intramuscularly, in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1562902A) (adjuvanted or not); Biological: Fluarix
- GSK1562902A 3 Group (Experimental): Subjects aged 61 years or older at the time of first vaccination received 2 doses of GSK1562902A adjuvanted vaccine at Days 0 and 21. The vaccine was administered in the deltoid region of each arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1562902A) (adjuvanted or not); Biological: Fluarix
- GSK1562902A 4 Group (Experimental): Subjects aged 61 years or older at the time of first vaccination received 2 doses of GSK1562902A non-adjuvanted vaccine at Days 0 and 21. The vaccine was administered in the deltoid region of each arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1562902A) (adjuvanted or not); Biological: Fluarix

INTERVENTIONS:
Biological: Pandemic influenza vaccine (GSK1562902A) (adjuvanted or not) — intramuscular injection
Biological: Fluarix — Intramuscular injection. All subjects not vaccinated with an influenza vaccine for the 2006-2007 season received Fluarix NH 2006/2007 (i.e. interpandemic GSK's influenza vaccine) at least 3 weeks before administration of the first dose of H5N1 vaccine.

SUMMARY:
The present study is designed to evaluate the immunogenicity and safety of a single or double dose of the pandemic influenza candidate vaccine (GSK1562902A), administered following a two-administration schedule (21 days apart) in adults over 60 years of age. The persistence of influenza antibodies will also be evaluated 24 months after vaccination.

DETAILED DESCRIPTION:
The present study is designed to evaluate the immunogenicity and safety of a single or double dose of the candidate vaccine in healthy elderly persons. The candidate vaccine will be administered following a two-administration schedule (21 days apart) in adults over 60 years of age. The persistence of H5N1 influenza antibodies will also be evaluated up to two years after vaccination (neutralizing antibodies will only be evaluated in a subset of subjects in the adjuvanted groups). Single and double dose of H5N1 vaccine non-adjuvanted vaccine will be used as comparator.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged 61 years or above at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects or subjects with well controlled underlying disease.

Exclusion Criteria:

* Administration of the licensed MF59-containing vaccines, e.g. Fluad™ or Addigrip™ or virosome-based influenza vaccines such as Inflexal V™, InfectoVac Flu™ or Invivac™ during the 2006-2007 influenza season.
* Administration of licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study.
* Planned administration of a vaccine not foreseen by the study protocol up to 30 days after the second vaccination with H5N1 vaccine.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of chronic alcohol consumption and/or drug abuse.
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (including egg and thiomersal allergy).
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Acute disease at the time of enrolment.
* Serious chronic disease including any medically significant chronic pulmonary, cardiovascular, renal, neurological, psychiatric or metabolic disorder, as determined by medical history and physical examination.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first vaccination or during the study.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to the first vaccination, or planned use during the study period.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2006-11-17 (Actual); Primary Completion 2009-09-14 (Actual); Study Completion 2009-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Belgium (7):
  - GSK Investigational Site, Dour
  - GSK Investigational Site, Gozée
  - GSK Investigational Site, Libramont
  - GSK Investigational Site, Mont-Godinne
  - GSK Investigational Site, Sprimont
  - GSK Investigational Site, Tessenderlo
  - GSK Investigational Site, Watermael-Boitsfort
- Italy (5):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monserrato Cagliari, Sardinia
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Ragusa, Sicily

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Gillard P, Giet D, Heijmans S, Drame M, Walravens K, Roman F. Long-term outcome of the humoral and cellular immune response of an H5N1 adjuvanted influenza vaccine in elderly persons: 2-year follow-up of a randomised open-label study. Trials. 2014 Oct 29;15:419. doi: 10.1186/1745-6215-15-419. PMID 25354581
- [Background] Heijmans S, De Meulemeester M, Reynders P, Giet D, Demanet E, Devresse PY, Icardi G, Drame M, Roman F, Gillard P. Immunogenicity profile of a 3.75-mug hemagglutinin pandemic rH5N1 split virion AS03A-adjuvanted vaccine in elderly persons: a randomized trial. J Infect Dis. 2011 Apr 15;203(8):1054-62. doi: 10.1093/infdis/jiq174. PMID 21450995
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 108251 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108251 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108251 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108251 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108251 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108251 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 108251 are summarised with studies 108252, 111275, and 111276 on the GSK Clinical Study Register.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects not previously vaccinated with an influenza vaccine for the 2006-2007 season were administered FluarixTM vaccine intramuscularly at least 3 weeks before administration of the first dose(s) of the GSK1562902A vaccine.
Groups:
- GSK1562902A 3 Group: Subjects aged 61 years or older at the time of first vaccination received 2 doses of GSK1562902A adjuvanted vaccine at Days 0 and 21. The vaccine was administered in deltoid region of each arm.
- GSK1562902A 4 Group: Subjects aged 61 years or older at the time of first vaccination received 2 doses of GSK1562902A non-adjuvanted vaccine at Days 0 and 21. The vaccine was administered in deltoid region of each arm.
Period: Month 0 (Day 0)
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Started | 165 | 61 | 159 | 52
Completed | 158 | 56 | 153 | 48
Not Completed | 7 | 5 | 6 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 3 | 1
Not completed — Other | 4 | 1 | 3 | 3
Period: Month 6 (Day 180)
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Started | 164 | 58 | 158 | 51
Completed | 162 | 55 | 153 | 51
Not Completed | 2 | 3 | 5 | 0
Not completed — Adverse Event | 0 | 3 | 2 | 0
Not completed — Other | 2 | 0 | 3 | 0
Period: Month 12 (Day 360)
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Started | 130 | 48 | 125 | 42
Completed | 130 | 48 | 125 | 42
Not Completed | 0 | 0 | 0 | 0
Period: Month 24 (Day 720)
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Started | 122 | 45 | 117 | 36
Completed | 122 | 45 | 117 | 36
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group | Total
Number analyzed (Participants) | 165 | 61 | 159 | 52 | 437
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.7 (6.33) | 69.9 (6.38) | 69.7 (6.51) | 70.8 (7.35) | 70.0 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 28 | 77 | 23 | 200
  Male | 93 | 33 | 82 | 29 | 237

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Two Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1). The reference seropositivity cut-off value was ≥ 1:10.
Time Frame: At Days 0, 21 and 42
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning Immunogenicity outcomes variables were available and for whom assay results were available for antibodies against at least one study vaccine component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 152 | 54 | 145 | 44
Titer
  A/Vietnam/1194/2004, Day 0 | 11.3 [9.2 to 13.9] | 9.7 [7.3 to 13.0] | 10.2 [8.4 to 12.5] | 8.8 [6.6 to 11.8]
  A/Vietnam/1194/2004, Day 21 | 50.0 [38.1 to 65.6] | 16.8 [11.7 to 24.0] | 69.4 [52.1 to 92.3] | 20.8 [13.0 to 33.3]
  A/Vietnam/1194/2004, Day 42 | 126.8 [99.4 to 161.7] | 22.7 [15.1 to 34.1] | 237.3 [191.9 to 293.6] | 25.3 [16.0 to 40.1]
  A/Indonezia/5/2005, Day 0 | 5.1 [5.0 to 5.1] | 5.2 [4.9 to 5.5] | 5.1 [5.0 to 5.2] | 5.0 [5.0 to 5.0]
  A/Indonezia/5/2005, Day 21 | 6.9 [6.2 to 7.7] | 5.3 [4.8 to 5.9] | 8.6 [7.3 to 10.1] | 5.6 [5.0 to 6.3]
  A/Indonezia/5/2005, Day 42 | 13.7 [11.3 to 16.4] | 6.1 [5.1 to 7.4] | 24.4 [19.9 to 30.0] | 6.3 [5.2 to 7.6]

2. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease.
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: At Days 21 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 152 | 54 | 145 | 44
Fold
  A/Vietnam/1994/2004, Day 21 | 4.4 [3.5 to 5.5] | 1.7 [1.3 to 2.3] | 6.8 [5.3 to 8.6] | 2.4 [1.7 to 3.4]
  A/Vietnam/1994/2004, Day 42 | 11.2 [8.9 to 14.1] | 2.3 [1.6 to 3.3] | 23.2 [18.5 to 29.0] | 2.9 [2.0 to 4.1]
  A/Indonezia/5/2005, Day 21 | 1.4 [1.2 to 1.5] | 1.0 [0.9 to 1.1] | 1.7 [1.4 to 2.0] | 1.1 [1.0 to 1.3]
  A/Indonezia/5/2005, Day 42 | 2.7 [2.2 to 3.2] | 1.2 [1.0 to 1.4] | 4.8 [3.9 to 5.9] | 1.3 [1.0 to 1.5]

3. Primary Outcome: Number of Seroprotected Subjects Against 2 Strains of Influenza Disease
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 152 | 54 | 145 | 44
Subjects
  A/Vietnam/1194/2004, Day 0 | 28 | 7 | 23 | 2
  A/Vietnam/1194/2004, Day 21 | 93 | 15 | 90 | 15
  A/Vietnam/1194/2004, Day 42 | 127 | 19 | 139 | 17
  A/Indonezia/5/2005, Day 0 | 0 | 0 | 0 | 0
  A/Indonezia/5/2005, Day 21 | 5 | 1 | 13 | 1
  A/Indonezia/5/2005, Day 42 | 35 | 2 | 59 | 2

4. Primary Outcome: Neutralizing Antibody Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Two Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1). The reference seropositivity cut-off value was ≥ 1:28. This outcome only covers results from the adjuvanted groups.
Time Frame: At Days 0 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 1 Group | GSK1562902A 3 Group
Number analyzed (Participants) | 87 | 82
Titer
  A/Vietnam/1194/2004, Day 0 | 121.1 [94.6 to 154.9] | 112.5 [90.7 to 139.5]
  A/Vietnam/1194/2004, Day 42 | 447.3 [359.3 to 557.0] | 595.8 [487.7 to 727.8]
  A/Indonesia/5/2005, Day 0 | 44.2 [36.0 to 54.1] | 39.7 [32.0 to 49.3]
  A/Indonesia/5/2005, Day 42 | 107.5 [88.9 to 130.0] | 169.6 [144.7 to 198.9]

5. Primary Outcome: Number of Seroconverted Subjects Against 2 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: At Days 21 and 42
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 152 | 54 | 145 | 44
Subjects
  A/Vietnam/1194/2004, Day 21 (N=152,54,145,44) | 69 | 8 | 76 | 8
  A/Vietnam/1194/2004, Day 42 (N=152,54,145,44) | 110 | 12 | 128 | 10
  A/Indonezia/5/2005, Day 21 (N=152,54,145,44) | 5 | 1 | 13 | 1
  A/Indonezia/5/2005, Day 42 (N=152,54,145,44) | 35 | 2 | 58 | 2

6. Primary Outcome: Number of Seroconverted Subjects for Neutralizing Antibody Response Against 2 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1). This outcome only covers results from the adjuvanted groups.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 3 Group
Number analyzed (Participants) | 87 | 82
Subjects
  A/Vitenam/1194/2004, Day 42 | 39 | 46
  A/Indonesia/5/2005, Day 42 | 25 | 40

7. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Two Strains of Influenza Disease.
Description: as for outcome 1
Time Frame: At Day 180
Population: The analysis was performed on the According-To-Protocol cohort for persistence, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol procedures during the entire study period and for whom assay results for antibodies against at least one study vaccine antigen component were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- GSK1562902A 2 Group: GSK1562902A 2 Group Subjects aged 61 years or older at the time of first vaccination received 1 dose of GSK1562902A non-adjuvanted vaccine at Day 0. The vaccine was administered intramuscularly, in the deltoid region of the non-dominant arm.
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 140 | 50 | 131 | 44
Titers
  A/Vietnam/1194/2004 | 38.5 [30.0 to 49.5] | 16.3 [11.0 to 24.3] | 53.5 [41.9 to 68.4] | 13.1 [8.9 to 19.2]
  A/Indonezia/5/2005 | 6.6 [6.0 to 7.3] | 5.5 [4.8 to 6.4] | 8.6 [7.5 to 9.9] | 5.2 [4.8 to 5.5]

8. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Two Strains of Influenza Disease.
Description: as for outcome 1
Time Frame: At Month 12
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 112 | 45 | 106 | 35
Titer
  A/Vietnam/1194/2004 | 21.4 [16.4 to 28.0] | 13.3 [9.3 to 19.0] | 26.5 [20.3 to 34.6] | 11.4 [7.7 to 16.7]
  A/Indonezia/5/2005 | 9.8 [8.2 to 11.7] | 6.6 [5.5 to 7.9] | 13.1 [10.9 to 15.8] | 6.9 [5.4 to 8.9]

9. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Two Strains of Influenza Disease.
Description: as for outcome 1
Time Frame: At Month 24
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 86 | 37 | 81 | 24
Titer
  A/Vietnam/1194/2004 | 17.6 [13.7 to 22.5] | 12.3 [8.9 to 16.9] | 18.4 [14.2 to 23.8] | 9.8 [6.7 to 14.4]
  A/Indonezia/5/2005 | 7.0 [6.1 to 8.1] | 5.6 [4.9 to 6.4] | 7.3 [6.2 to 8.6] | 5.0 [5.0 to 5.0]

10. Primary Outcome: Number of Seroconverted Subjects Against 2 Strains of Influenza Disease.
Description: as for outcome 5
Time Frame: At Day 180
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 140 | 48 | 130 | 42
Subjects
  A/Vietnam/1194/2004 | 52 | 6 | 70 | 6
  A/Indonezia/5/2005 | 5 | 1 | 8 | 0

11. Primary Outcome: Number of Seroconverted Subjects Against 2 Strains of Influenza Disease.
Description: as for outcome 5
Time Frame: At Month 12
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 112 | 43 | 105 | 34
Subjects
  A/Vietnam/1194/2004 | 24 | 6 | 24 | 4
  A/Indonezia/5/2005 | 17 | 2 | 22 | 3

12. Primary Outcome: Number of Seroconverted Subjects Against 2 Strains of Influenza Disease.
Description: as for outcome 5
Time Frame: At Month 24
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 86 | 36 | 81 | 22
Subjects
  A/Vietnam/1194/2004 | 8 | 2 | 9 | 2
  A/Indonezia/5/2005 | 4 | 1 | 4 | 0

13. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease.
Description: as for outcome 2
Time Frame: At Day 180
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Fold
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 140 | 48 | 130 | 42
Fold
  A/Vietnam/1994/2004 | 3.3 [2.7 to 4.0] | 1.6 [1.2 to 2.2] | 5.4 [4.4 to 6.7] | 1.8 [1.3 to 2.4]
  A/Indonezia/5/2005 | 1.3 [1.2 to 1.4] | 1.1 [0.9 to 1.3] | 1.7 [1.5 to 1.9] | 1.0 [1.0 to 1.1]

14. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 2
Time Frame: At Month 12
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Fold
Groups:
- GSK1562902A 3 Group: GSK1562902A 3 Group Subjects aged 61 years or older at the time of first vaccination received 2 doses of GSK1562902A adjuvanted vaccine at Days 0 and 21. The vaccine was administered in deltoid region of each arm.
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 112 | 43 | 105 | 34
Fold
  A/Vietnam/1994/2004 | 1.8 [1.5 to 2.2] | 1.3 [1.0 to 1.7] | 2.5 [2.0 to 3.0] | 1.5 [1.1 to 2.1]
  A/Indonezia/5/2005 | 1.9 [1.6 to 2.3] | 1.3 [1.1 to 1.6] | 2.6 [2.2 to 3.1] | 1.4 [1.1 to 1.8]

15. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 2
Time Frame: At Month 24
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Fold
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 86 | 36 | 81 | 22
Fold
  A/Vietnam/1994/2004 | 1.5 [1.3 to 1.8] | 1.3 [0.9 to 1.7] | 1.9 [1.6 to 2.3] | 1.4 [1.0 to 2.1]
  A/Indonezia/5/2005 | 1.4 [1.2 to 1.6] | 1.1 [1.0 to 1.3] | 1.4 [1.2 to 1.7] | 1.0 [1.0 to 1.0]

16. Primary Outcome: Number of Seroprotected Subjects Against 2 Strains of Influenza Disease
Description: as for outcome 3
Time Frame: At Day 180
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 140 | 50 | 131 | 44
Subjects
  A/Vietnam/1194/2004 | 74 | 13 | 91 | 9
  A/Indonezia/5/2005 | 5 | 1 | 8 | 0

17. Primary Outcome: Number of Seroprotected Subjects Against 2 Strains of Influenza Disease
Description: as for outcome 3
Time Frame: At Month 12
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 112 | 45 | 106 | 35
Subjects
  A/Vietnam/1194/2004 | 49 | 11 | 45 | 7
  A/Indonezia/5/2005 | 17 | 2 | 22 | 3

18. Primary Outcome: Number of Seroprotected Subjects Against 2 Strains of Influenza Disease
Description: as for outcome 3
Time Frame: At Month 24
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 86 | 37 | 81 | 24
Subjects
  A/Vietnam/1194/2004 | 32 | 6 | 25 | 2
  A/Indonezia/5/2005 | 4 | 1 | 5 | 0

19. Primary Outcome: Number of Seroconverted Subjects for Neutralizing Antibody Response Against 2 Strains of Influenza Disease.
Description: as for outcome 6
Time Frame: At Day 180
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 3 Group
Number analyzed (Participants) | 76 | 73
Subjects
  A/Vietnam/1194/2004 | 16 | 21
  A/Indonesia/5/2005 | 20 | 32

20. Primary Outcome: Number of Seroconverted Subjects for Neutralizing Antibody Response Against 2 Strains of Influenza Disease.
Description: as for outcome 6
Time Frame: At Month 12
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 3 Group
Number analyzed (Participants) | 69 | 71
Subjects
  A/Vietnam/1194/2004 | 18 | 21
  A/Indonesia/5/2005 | 13 | 28

21. Primary Outcome: Number of Seroconverted Subjects for Neutralizing Antibody Response Against 2 Strains of Influenza Disease.
Description: as for outcome 6
Time Frame: At Month 24
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 3 Group
Number analyzed (Participants) | 49 | 54
Subjects
  A/Vietnam/1194/2004 | 18 | 22
  A/Indonesia/5/2005 | 6 | 16

22. Primary Outcome: Neutralizing Antibody Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Two Strains of Influenza Disease.
Description: as for outcome 4
Time Frame: At Month 12
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 1 Group | GSK1562902A 3 Group
Number analyzed (Participants) | 69 | 71
Titer
  A/Vietnam/1194/2004 | 274.7 [213.4 to 353.5] | 268.8 [211.4 to 341.8]
  A/Indonesia/5/2005 | 82.5 [63.0 to 107.9] | 119.8 [94.0 to 152.7]

23. Primary Outcome: Neutralizing Antibody Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Two Strains of Influenza Disease.
Description: as for outcome 4
Time Frame: At Month 24
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 1 Group | GSK1562902A 3 Group
Number analyzed (Participants) | 76 | 73
Titer
  A/Vietnam/1194/2004 | 391.0 [295.5 to 517.5] | 382.8 [317.4 to 461.6]
  A/Indonesia/5/2005 | 75.4 [57.2 to 99.4] | 84.9 [67.0 to 107.6]

24. Primary Outcome: Neutralizing Antibody Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Two Strains of Influenza Disease.
Description: as for outcome 4
Time Frame: At Day 180
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 1 Group | GSK1562902A 3 Group
Number analyzed (Participants) | 76 | 73
Titer
  A/Vietnam/1194/2004 | 218.2 [172.4 to 276.2] | 260.9 [207.7 to 327.8]
  A/Indonesia/5/2005 | 97.8 [82.0 to 116.5] | 134.5 [113.4 to 159.7]

25. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration. Note: No AESIs were reported during the entire study period.
Time Frame: During the entire study period (Day 0 to Month 24)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available, on a subset of subjects enrolled for this study in Belgium.
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 ecchymosis/induration/redness/swelling = ecchymosis/induration/redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day follow-up period (Days 0 to 6) after any vaccination
Population: The analysis was based on the Total Vaccinated Cohort, which included all subjects with at least one documented dose, for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 164 | 61 | 159 | 51
Subjects
  Ecchymosis | 1 | 0 | 5 | 1
  Induration | 10 | 0 | 15 | 0
  Pain | 69 | 6 | 75 | 3
  Redness | 19 | 0 | 30 | 1
  Swelling | 19 | 0 | 15 | 0
  Ecchymosis >100mm | 0 | 0 | 0 | 0
  Induration >100mm | 0 | 0 | 0 | 0
  Grade 3 Pain | 0 | 0 | 2 | 0
  Redness >100mm | 0 | 0 | 1 | 0
  Swelling >100mm | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Subjects With Abnormalities in Assessed Biochemical and Hematological Laboratory Parameters.
Description: Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), basophils (BAS), creatinine phosphokinase (CRPH), creatinine (CREA), eosinophils (EOS), haemoglobin (HEM), lactate dehydrogenase (LDE), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC), urea (URE) and white blood cells (WBC). Per parameter and range, it was assessed whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for ALT, AST, BAS, CREA and CRPH.
Time Frame: At Days 0, 2, 21 and 23
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 165 | 61 | 159 | 52
Subjects
  ALT, PRE (Day 0), Below (N=165,61,159,52) | 0 | 0 | 1 | 0
  ALT, PRE (Day 0), Normal (N=165,61,159,52) | 152 | 58 | 152 | 47
  ALT, PRE (Day 0), Above (N=165,61,159.52) | 13 | 3 | 6 | 5
  ALT, POST (Day2), Below (N=165,61,158,52) | 0 | 0 | 1 | 0
  ALT, POST (Day2), Normal (N=165,61,158,52) | 152 | 59 | 151 | 48
  ALT, POST (Day 2), Above (N=165,61,158,52) | 13 | 2 | 6 | 4
  ALT, POST (Day 21), Below (N=163,57,156,52) | 0 | 0 | 1 | 0
  ALT, POST (Day 21), Normal (N=163,57,156,52) | 153 | 54 | 144 | 48
  ALT, POST (Day 21), Above (N=163,57,156,52) | 10 | 3 | 11 | 4
  ALT, POST (Day23), Below (N=163,57,155,52) | 0 | 0 | 1 | 0
  ALT, POST (Day 23), Normal (N=163,57,155,52) | 152 | 55 | 146 | 49
  ALT, POST (Day 23), Above (N=163,57,155,52) | 11 | 2 | 8 | 3
  AST, PRE (Day 0), Below (N=165,61,159,52) | 0 | 0 | 0 | 0
  AST, PRE (Day 0), Normal (N=165,61,159,52) | 154 | 57 | 150 | 48
  AST, PRE (Day 0), Above (N=165,61,159,52) | 11 | 4 | 9 | 4
  AST, POST (Day 2), Below (N=165,61,158,52) | 0 | 0 | 0 | 0
  AST, POST (Day 2), Normal (N=165,61,158,52) | 154 | 59 | 152 | 49
  AST, POST (Day 2), Above (N=165,61,158,52) | 11 | 2 | 6 | 3
  AST, POST (Day 21), Below (N=163,57,156,52) | 0 | 0 | 0 | 0
  AST, POST (Day 21), Normal (N=163,57,156,52) | 154 | 51 | 146 | 47
  AST, POST (Day 21), Above (N=163,57,156,52) | 9 | 6 | 10 | 5
  AST, POST (Day 23), Below (N=163,57,155,52) | 0 | 0 | 0 | 0
  AST, POST (Day 23), Normal (N=163,57,155,52) | 153 | 54 | 149 | 47
  AST, POST (Day 23), Above (N=163,57,155,52) | 10 | 3 | 6 | 5
  BAS, PRE (Day 0), Below (N=163,61,159,52) | 0 | 0 | 0 | 0
  BAS, PRE (Day 0), Normal (N=163,61,159,52) | 163 | 61 | 159 | 52
  BAS, PRE (Day 0), Above (N=163,61,159,52) | 0 | 0 | 0 | 0
  BAS, POST (Day 2), Below (N=165,61,158,52) | 0 | 0 | 0 | 0
  BAS, POST (Day 2), Normal (N=165,61,158,52) | 164 | 61 | 158 | 52
  BAS, POST (Day 2), Above (N=165,61,158,52) | 1 | 0 | 0 | 0
  BAS, POST (Day 21), Below (N=163,57,155,52) | 0 | 0 | 0 | 0
  BAS, POST (Day 21), Normal (N=163,57,155,52) | 163 | 57 | 155 | 52
  BAS, POST (Day 21), Above (N=163,57,155,52) | 0 | 0 | 0 | 0
  BAS, POST (Day 23), Below (N=163, 57,155,51) | 0 | 0 | 0 | 0
  BAS, POST (Day 23), Below (N=163,57,155,51) | 163 | 57 | 155 | 51
  BAS, POST (Day 23), Above (N=163,57,155,51) | 0 | 0 | 0 | 0
  CREA, PRE (Day 0), Below (N=165,61,159,52) | 0 | 1 | 0 | 0
  CREA, PRE (Day 0), Normal (N=165,61,159,52) | 144 | 54 | 148 | 43
  CREA, PRE (Day 0), Above (N=165,61,159,52) | 21 | 6 | 11 | 9
  CREA, POST (Day 2), Below (N=165,61,158,51) | 1 | 0 | 1 | 0
  CREA, POST (Day 2), Normal (N=165,61,158,51) | 144 | 55 | 146 | 42
  CREA, POST (Day 2), Above (N=165,61,158,51) | 20 | 6 | 11 | 9
  CREA, POST (Day 21), Below (N=163,57,156,52) | 0 | 0 | 1 | 0
  CREA, POST (Day 21), Normal (N=163,57,156,52) | 134 | 51 | 142 | 42
  CREA, POST (Day 21), Above (N=163,57,156,52) | 29 | 6 | 13 | 10
  CREA, POST (Day 23), Below (N=163,57,155,52) | 1 | 0 | 1 | 0
  CREA, POST (Day 23), Normal (N=163,57,155,52) | 142 | 49 | 139 | 45
  CREA, POST (Day 23), Above (N=163,57,155,52) | 20 | 8 | 15 | 7
  CRPH, PRE (Day 0), Below (N=165,60,158,52) | 0 | 0 | 0 | 0
  CRPH, PRE (Day 0), Normal (N=165,60,158,52) | 149 | 45 | 136 | 47
  CRPH, PRE (Day 0), Above (N=165,60,158,52) | 16 | 15 | 22 | 5
  CRPH, POST (Day 2), Below (N=165,61,158,52) | 0 | 0 | 1 | 0
  CRPH, POST (Day 2), Normal (N=165,61,158,52) | 150 | 49 | 141 | 44
  CRPH, POST (Day 2), Above (N=165,61,158,52) | 15 | 12 | 16 | 8
  CRPH, POST (Day 21), Below (N=163,57,156,52) | 1 | 0 | 0 | 0
  CRPH, POST (Day 21), Normal (N=163,57,156,52) | 140 | 45 | 130 | 45
  CRPH, POST (Day 21), Above (N=163,57,156,52) | 22 | 12 | 26 | 7
  CRPH, POST (Day 23), Below (N=163,57,155,52) | 0 | 0 | 0 | 0
  CRPH, POST (Day 23), Normal (N=163,57,155,52) | 146 | 49 | 136 | 44
  CRPH, POST (Day 23), Above (N=163,57,155,52) | 17 | 8 | 19 | 8

28. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Note: The study period was divided into 4 consecutive periods (Days 0-51, Days 52-180 [Month 6], Months 6-12 and Months 12-24), for which SAEs were collected.
Time Frame: During the entire study period (Day 0 to Month 24).
Population: The analysis was based on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 165 | 61 | 159 | 52
Subjects
  Subjects with SAEs Days 0-51 [N=165,61,159,52] | 1 | 1 | 1 | 1
  Subjects with SAEs Days 52-180 [N=164,58,158,51] | 5 | 3 | 5 | 0
  Subjects with SAEs Months 6-12 [N=130,48,125,42] | 4 | 0 | 3 | 2
  Subjects with SAEs Months 12-24 [N=122,45,117,36] | 9 | 7 | 7 | 2

29. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 21-day (Days 0-20) follow-up period after first vaccination and during the 30-day (Days 0-29) follow-up period after second vaccination
Population: as for outcome 28
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 165 | 61 | 159 | 52
Subjects
  Subjects with any AEs | 36 | 16 | 28 | 8
  Subjects with Grade 3 AEs | 5 | 2 | 3 | 1
  Subjects with related AEs | 9 | 2 | 10 | 1

30. Secondary Outcome: Number of Subjects With Abnormalities in Assessed Biochemical and Hematological Laboratory Parameters.
Description: Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), basophils (BAS), creatinine phosphokinase (CRPH), creatinine (CREA), eosinophils (EOS), haemoglobin (HEM), lactate dehydrogenase (LDE), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC), urea (URE) and white blood cells (WBC). Per parameter and range, it was assessed whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents EOS, HEM, LDE, LYM and MON results.
Time Frame: At Days 0, 2, 21 and 23.
Population: as for outcome 28
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 165 | 61 | 159 | 52
Subjects
  EOS, PRE (Day 0), Below (N=163,61,159,52) | 4 | 3 | 5 | 2
  EOS, PRE (Day 0), Normal (N=163,61,159,52) | 159 | 58 | 153 | 50
  EOS, PRE (Day 0), Above (N=163,61,159,52) | 0 | 0 | 1 | 0
  EOS, POST (Day 2), Below (N=165,61,158,52) | 4 | 3 | 5 | 3
  EOS, POST (Day 2), Normal (N=165,61,158,52) | 161 | 58 | 152 | 49
  EOS, POST (Day 2), Above (N=165,61,158,52) | 0 | 0 | 1 | 0
  EOS, POST (Day 21), Below (N=163,57,155,52) | 4 | 0 | 4 | 2
  EOS, POST (Day 21), Normal (N=163,57,155,52) | 158 | 57 | 150 | 50
  EOS, POST (Day 21), Above (N=163,57,155,52) | 1 | 0 | 1 | 0
  EOS, POST (Day 23), Below (N=163,57,155,51) | 4 | 0 | 4 | 2
  EOS, POST (Day 23), Normal (N=163,57,155,51) | 159 | 57 | 149 | 49
  EOS, POST (Day 23), Above (N=163,57,155,51) | 0 | 0 | 2 | 0
  HEM, PRE (Day 0), Below (N=163,61,159,52) | 11 | 3 | 14 | 3
  HEM, PRE (Day 0), Normal (N=163,61,159,52) | 137 | 50 | 130 | 43
  HEM, PRE (Day 0), Above (N=163,61,159,52) | 15 | 8 | 15 | 6
  HEM, POST (Day 2), Below (N=165,61,158,52) | 21 | 6 | 16 | 3
  HEM, POST (Day 2), Normal (N=165,61,158,52) | 139 | 53 | 135 | 47
  HEM, POST (Day 2), Above (N=165,61,158,52) | 5 | 2 | 7 | 2
  HEM, POST (Day 21), Below (N=163,57,155,52) | 13 | 2 | 15 | 4
  HEM, POST (Day 21), Normal (N=163,57,155,52) | 144 | 53 | 130 | 44
  HEM, POST (Day 21), Above (N=163,57,155,52) | 6 | 2 | 10 | 4
  HEM, POST (Day 23), Below (N=163,57,155,52) | 20 | 3 | 17 | 5
  HEM, POST (Day 23), Normal (N=163,57,155,52) | 139 | 54 | 133 | 44
  HEM, POST (Day 23), Above (N=163,57,155,52) | 4 | 0 | 5 | 3
  LDE, PRE (Day 0), Below (N=164,61,156,52) | 1 | 2 | 2 | 0
  LDE, PRE (Day 0), Normal (N=164,61,156,52) | 147 | 51 | 136 | 49
  LDE, PRE (Day 0), Above (N=164,61,156,52) | 16 | 8 | 18 | 3
  LDE, POST (Day 2), Below (N=165,61,158,52) | 2 | 1 | 2 | 0
  LDE, PRE (Day 2), Normal (N=165,61,158,52) | 148 | 56 | 144 | 45
  LDE, PRE (Day 2), Above (N=165,61,158,52) | 15 | 4 | 12 | 7
  LDE, POST (Day 21), Below (N=162,57,156,52) | 0 | 1 | 1 | 0
  LDE, POST (Day 21), Normal (N=162,57,156,52) | 151 | 44 | 142 | 48
  LDE, POST (Day 21), Above (N=162,57,156,52) | 11 | 12 | 13 | 4
  LDE, POST (Day 23), Below (N=163,57,155,52) | 4 | 1 | 2 | 0
  LDE, POST (Day 23), Normal (N=163,57,155,52) | 147 | 54 | 141 | 50
  LDE, POST (Day 23), Above (N=163,57,155,52) | 12 | 2 | 12 | 2
  LYM, PRE (Day 0), Below (N=163,61,159,52) | 145 | 53 | 137 | 45
  LYM, PRE (Day 0), Normal (N=163,61,159,52) | 18 | 8 | 22 | 7
  LYM, PRE (Day 0), Above (N=163,61,159,52) | 0 | 0 | 0 | 0
  LYM, POST (Day 2), Below (N=165,61,158,52) | 148 | 53 | 136 | 46
  LYM, POST (Day 2), Normal (N=165,61,158,52) | 17 | 8 | 22 | 6
  LYM, POST (Day 2), Above (N=165,61,158,52) | 0 | 0 | 0 | 0
  LYM, POST (Day 21), Below (N=163,57,155,52) | 144 | 52 | 135 | 45
  LYM, POST (Day 21), Normal (N=163,57,155,52) | 19 | 5 | 20 | 7
  LYM, POST (Day 21), Above (N=163,57,155,52) | 0 | 0 | 0 | 0
  LYM, POST (Day 23), Below (N=163,57,155,51) | 145 | 52 | 135 | 44
  LYM, POST (Day 23), Normal (N=163,57,155,51) | 17 | 5 | 20 | 7
  LYM, POST (Day 23), Above (N=163,57,155,51) | 1 | 0 | 0 | 0
  MON, PRE (Day 0), Below (N=163,61,159,52) | 143 | 52 | 136 | 45
  MON, PRE (Day 0), Normal (N=163,61,159,52) | 20 | 9 | 23 | 7
  MON, PRE (Day 0), Above (N=163,61,159,52) | 0 | 0 | 0 | 0
  MON, POST (Day 2), Below (N=165,61,158,52) | 143 | 53 | 134 | 45
  MON, POST (Day 2), Normal (N=165,61,158,52) | 21 | 8 | 24 | 7
  MON, POST (Day 2), Above (N=165,61,158,52) | 1 | 0 | 0 | 0
  MON, POST (Day 21), Below (N=163,57,155,52) | 140 | 52 | 134 | 45
  MON, POST (Day 21), Normal (N=163,57,155,52) | 23 | 5 | 21 | 7
  MON, POST (Day 21), Above (N=163,57,155,52) | 0 | 0 | 0 | 0
  MON, POST (Day 23), Below (N=163,57,155,51) | 141 | 52 | 134 | 44
  MON, POST (Day 23), Normal (N=163,57,155,51) | 19 | 5 | 17 | 7
  MON, POST (Day 23), Above (N=163,57,155,51) | 3 | 0 | 4 | 0

31. Secondary Outcome: Geometric Mean of Influenza-specific Cluster of Differentiation (CD) 4/CD8 T-cells.
Description: The geometric mean was calculated for cluster of differentiation (CD) 4/CD 8 T-cells (per million) producing at least one cytokine beside either of the following: CD40 ligand [CD40L], interleukin-2 [IL-2], tumor necrosis factor-alpha [TNF-α] or interferon-gamma [IFN-γ].
Time Frame: At Month 12
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: Cells
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 90 | 41 | 91 | 30
Cells
  CD4 All doubles | 898.52 (1050.39) | 693.48 (668.33) | 1170.36 (1021.43) | 869.43 (632.5)
  CD4-CD40L | 934.35 (1020.83) | 675.52 (655.85) | 1146.47 (1002.22) | 850.8 (612.75)
  CD4-IL-2 | 902.69 (1006.77) | 623.44 (623.44) | 1118.63 (973.32) | 798.58 (598.14)
  CD4-INF-g | 442.66 (743.99) | 442.16 (419.92) | 586.6 (577.71) | 542.62 (471.58)
  CD4-TNF-a | 678.6 (870.28) | 515.7 (484.61) | 884.64 (847.51) | 647.75 (528.32)
  CD8 All doubles | 34.28 (275.22) | 29.42 (283.23) | 27.88 (261.68) | 34.21 (838.37)
  CD8-CD40L | 2.08 (28.46) | 2.22 (20.24) | 2.99 (28.9) | 2.48 (31.11)
  CD8-IL-2 | 18.84 (167.58) | 24.72 (153.94) | 19.95 (164.36) | 28.85 (598.65)
  CD8-INF-g | 29.13 (271.12) | 24.45 (285.49) | 20.75 (260.19) | 32.99 (829.25)
  CD8-TNF-a | 35.67 (251.66) | 32.59 (230.03) | 28.15 (246.49) | 31.35 (595.41)

32. Secondary Outcome: Geometric Mean of Influenza-specific Cluster of Differentiation (CD) 4/CD8 T-cells.
Description: as for outcome 31
Time Frame: At Month 24
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: Cells
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 73 | 34 | 72 | 22
Cells
  CD4 All doubles [N=73,34,72,22] | 779.93 (771.46) | 569.84 (1058.95) | 1126.86 (1375.31) | 832.74 (908.25)
  CD4-CD40L [N=73,34,72,22] | 710.53 (712.25) | 454.56 (1060.83) | 1041.16 (1356.01) | 740.77 (820.93)
  CD4-IL-2 [N=73,34,72,22] | 769.56 (718.28) | 509.21 (1039.78) | 1043.95 (1333.41) | 783.88 (868.28)
  CD4-INF-g [N=73,34,72,22] | 455.05 (608.16) | 391.45 (923.81) | 651.02 (947.13) | 563.18 (849.25)
  CD4-TNF-a [N=73,34,72,22] | 500.82 (555.63) | 374.53 (962.01) | 806.94 (1012.4) | 598.88 (860.46)
  CD8 All doubles [N=73,33,72,22] | 8.05 (94.19) | 8.06 (60.49) | 21.67 (258.83) | 14.92 (381.27)
  CD8-CD40L [N=73,33,72,22] | 1.94 (29.28) | 2.65 (33.03) | 2.58 (32.7) | 1.48 (18.2)
  CD8-IL-2 [N=73,33,72,22] | 5.04 (65.04) | 4.16 (69.59) | 8.16 (181.28) | 6.51 (310.91)
  CD8-INF-g [N=73,33,72,22] | 7.43 (93.13) | 9.05 (79.82) | 23.39 (257.7) | 12.47 (382.05)
  CD8-TNF-a [N=73,33,72,22] | 4.76 (65.03) | 4.05 (51.49) | 17.22 (231.77) | 15.3 (325.83)

33. Secondary Outcome: Number of Subjects With Abnormalities in Assessed Biochemical and Hematological Laboratory Parameters.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (HEM), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Per parameter and range, it was assessed whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents NEU, PLA, RBC, URE and WBC results.
Time Frame: At Days 0, 2, 21 and 23.
Population: as for outcome 28
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 165 | 61 | 159 | 52
Subjects
  NEU, PRE (Day 0), Below (N=163,61,158,52) | 148 | 55 | 141 | 47
  NEU, PRE (Day 0), Normal (N=163,61,158,52) | 13 | 5 | 17 | 5
  NEU, PRE (Day 0), Above (N=163,61,158,52) | 2 | 1 | 0 | 0
  NEU, POST (Day 2), Below (N=165,61,158,52) | 149 | 55 | 141 | 47
  NEU, POST (Day 2), Normal (N=165,61,158,52) | 13 | 6 | 17 | 4
  NEU, POST (Day 2), Above (N=165,61,158,52) | 3 | 0 | 0 | 1
  NEU, POST (Day 21), Below (N=163,57,155,52) | 147 | 52 | 138 | 47
  NEU, POST (Day 21), Normal (N=163,57,155,52) | 14 | 4 | 15 | 4
  NEU, POST (Day 21), Above (N=163,57,155,52) | 2 | 1 | 2 | 1
  NEU, POST (Day 23), Below (N=163,57,155,51) | 148 | 52 | 138 | 46
  NEU, POST (Day 23), Normal (N=163,57,155,51) | 14 | 4 | 17 | 5
  NEU, POST (Day 23), Above (N=163,57,155,51) | 1 | 1 | 0 | 0
  PLA, PRE (Day 0), Below (N=163,61,159,52) | 4 | 4 | 3 | 2
  PLA, PRE (Day 0), Normal (N=163,61,159,52) | 145 | 51 | 148 | 46
  PLA, PRE (Day 0), Above (N=163,61,159,52) | 14 | 6 | 8 | 4
  PLA, POST (Day 2), Below (N=165,61,158,52) | 2 | 2 | 4 | 2
  PLA, POST (Day 2), Normal (N=165,61,158,52) | 152 | 51 | 147 | 45
  PLA, POST (Day 2), Above (N=165,61,158,52) | 11 | 8 | 7 | 5
  PLA, POST (Day 21), Below (N=163,57,155,52) | 3 | 6 | 4 | 1
  PLA, POST (Day 21), Normal (N=163,57,155,52) | 147 | 49 | 145 | 46
  PLA, POST (Day 21), Above (N=163,57,155,52) | 13 | 2 | 6 | 5
  PLA, POST (Day 23), Below (N=163,57,155,52) | 2 | 3 | 2 | 0
  PLA, POST (Day 23), Normal (N=163,57,155,52) | 150 | 52 | 147 | 48
  PLA, POST (Day 23), Above (N=163,57,155,52) | 11 | 2 | 6 | 4
  RBC, PRE (Day 0), Below (N=163,61,159,52) | 21 | 5 | 21 | 5
  RBC, PRE (Day 0), Normal (N=163,61,159,52) | 132 | 54 | 125 | 42
  RBC, PRE (Day 0), Above (N=163,61,159,52) | 10 | 2 | 13 | 5
  RBC, POST (Day 2), Below (N=165,61,158,52) | 25 | 8 | 20 | 7
  RBC, POST (Day 2), Normal (N=165,61,158,52) | 134 | 52 | 133 | 43
  RBC, POST (Day 2), Above (N=165,61,158,52) | 6 | 1 | 5 | 2
  RBC, POST (Day 21), Below (N=163,57,155,52) | 24 | 6 | 20 | 7
  RBC, POST (Day 21), Normal (N=163,57,155,52) | 133 | 47 | 127 | 42
  RBC, POST (Day 21), Above(N=163,57,155,52) | 6 | 4 | 8 | 3
  RBC, POST (Day23), Below (N=163,57,155,52) | 33 | 8 | 19 | 8
  RBC, POST (Day23), Normal (N=163,57,155,52) | 127 | 47 | 134 | 43
  RBC, POST (Day23), Above (N=163,57,155,52) | 3 | 2 | 2 | 1
  URE, PRE (Day 0), Below (N=165,61,159,52) | 0 | 0 | 4 | 0
  URE, PRE (Day 0), Normal (N=165,61,159,52) | 90 | 36 | 101 | 34
  URE, PRE (Day 0), Above (N=165,61,159,52) | 75 | 25 | 54 | 18
  URE, POST (Day 2), Below (N=164,61,158,52) | 1 | 0 | 4 | 0
  URE, POST (Day 2), Normal (N=164,61,158,52) | 96 | 38 | 114 | 32
  URE, POST (Day 2), Above (N=164,61,158,52) | 67 | 23 | 40 | 20
  URE, POST (Day 21), Below (N=163,57,156,52) | 0 | 0 | 3 | 0
  URE, POST (Day 21), Normal (N=163,57,156,52) | 91 | 30 | 100 | 32
  URE, POST (Day 21), Above (N=163,57,156,52) | 72 | 27 | 53 | 20
  URE, POST (Day 23), Below (N=163,57,155,52) | 0 | 0 | 2 | 0
  URE, POST (Day 23), Normal (N=163,57,155,52) | 105 | 36 | 106 | 36
  URE, POST (Day 23), Above (N=163,57,155,52) | 58 | 21 | 47 | 16
  WBC, PRE (Day 0), Below (N=163,61,159,52) | 5 | 2 | 3 | 3
  WBC, PRE (Day 0), Normal (N=163,61,159,52) | 152 | 56 | 155 | 45
  WBC, PRE (Day 0), Above (N=163,61,159,52) | 6 | 3 | 1 | 4
  WBC, POST (Day 2), Below (N=165,61,158,52) | 4 | 2 | 4 | 3
  WBC, POST (Day 2), Normal (N=165,61,158,52) | 152 | 56 | 152 | 47
  WBC, POST (Day 2), Above (N=165,61,158,52) | 9 | 3 | 2 | 2
  WBC, POST (Day 21), Below (N=163,57,155,52) | 4 | 2 | 3 | 3
  WBC, POST (Day 21), Normal (N=163,57,155,52) | 150 | 53 | 149 | 49
  WBC, POST (Day 21), Above (N=163,57,155,52) | 9 | 2 | 3 | 0
  WBC, POST (Day 23), Below (N=163,57,155,52) | 6 | 4 | 7 | 3
  WBC, POST (Day 23), Normal (N=163,57,155,52) | 145 | 49 | 148 | 47
  WBC, POST (Day 23), Above (N=163,57,155,52) | 12 | 4 | 0 | 2

34. Secondary Outcome: Geometric Mean of Influenza-specific Cluster of Differentiation (CD) 4/CD8 T-cells.
Description: The geometric mean was calculated for cluster of differentiation (CD) 4/CD 8 T-cells (per million) producing at least one cytokine beside either of the following: CD40 ligand [CD40L], interleukin-2 [IL-2], interferon gamma [INF-g] and tumor necrosis factor-alpha [TNF-α].
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Cells
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 129 | 44 | 122 | 40
Cells
  CD4 All doubles, Day 0 [N=129,44,122,40] | 393.71 (590.66) | 494.27 (518.93) | 495.77 (606.84) | 545.37 (820.30)
  CD4-CD40L, Day 0 [N=129,44,122,40] | 388.69 (571.91) | 461.29 (513.70) | 485.71 (594.88) | 540.73 (771.32)
  CD4-IL-2, Day 0 [N=129,44,122,40] | 376.03 (545.75) | 448.43 (500.03) | 461.23 (552.91) | 510.47 (700.70)
  CD4-INF-g, Day 0 [N=129,44,122,40] | 270.99 (500.13) | 322.17 (349.01) | 343.35 (549.24) | 371.67 (695.33)
  CD4-TNF-a, Day 0 [N=129,44,122,40] | 310.91 (486.27) | 369.54 (427.12) | 358.27 (538.07) | 382.79 (641.28)
  CD4 All doubles, Day 21 [N=112,42,110,34] | 1407.29 (1354.44) | 943.54 (1034.54) | 1793.92 (1867.92) | 1284.19 (1058.55)
  CD4-CD40L, Day 21 [N=112,42,110,34] | 1374.26 (1304.02) | 944.17 (1015.89) | 1731.58 (1828.74) | 1230.48 (989.52)
  CD4-IL-2, Day 21 [N=112,42,110,34] | 1318.03 (1250.79) | 868.24 (967.47) | 1651.88 (1776.72) | 1178.95 (1001.08)
  CD4-INF-g, Day 21 [N=112,42,110,34] | 685.44 (884.75) | 579.45 (828.17) | 997.15 (1023.96) | 852.75 (823.22)
  CD4-TNF-a, Day 21 [N=112,42,110,34] | 932.64 (974.72) | 708.15 (915.15) | 1207.95 (1527.86) | 910.69 (861.04)
  CD4 All doubles, Day 42 [N=120,43,118,30] | 2260.19 (2242.14) | 920.9 (745.36) | 3049.03 (4208.17) | 1316.8 (1060.97)
  CD4-CD40L, Day 42 [N=120,43,118,30] | 2198.66 (2165.46) | 944.59 (728.39) | 2971.34 (4076.52) | 1254.99 (974.2)
  CD4-IL-2, Day 42 [N=120,43,118,30] | 2086.84 (2086.66) | 854.9 (727.62) | 2762.65 (3720.42) | 1242.26 (976.18)
  CD4-INF-g, Day 42 [N=120,43,118,30] | 1123.16 (1356.18) | 671.86 (552.02) | 1535.37 (2864.48) | 828.99 (732.58)
  CD4-TNF-a, Day 42 [N=120,43,118,30] | 1595.64 (1798.95) | 701.35 (691.26) | 2170.46 (3380.48) | 918.5 (822.2)
  CD8 All doubles, Day 0 [N=129,44,121,40] | 83.30 (407.94) | 52.25 (497.68) | 71.93 (626.44) | 94.74 (1903.91)
  CD8-CD40L, Day 0 [N=129,44,121,40] | 3.37 (52.35) | 2.94 (34.07) | 3.58 (48.88) | 4.30 (322.83)
  CD8-IL-2, Day 0 [N=129,44,121,40] | 53.90 (241.03) | 43.45 (334.22) | 59.70 (340.60) | 56.29 (1426.27)
  CD8-INF-g, Day 0 [N=129,44,121,40] | 83.14 (394.32) | 44.71 (489.55) | 80.54 (618.55) | 98.30 (1888.61)
  CD8-TNF-a, Day 0 [N=129,44,121,40] | 63.19 (355.75) | 36.83 (414.08) | 45.34 (573.91) | 82.77 (1532.47)
  CD8 All doubles, Day 21 [N=111,41,109,34] | 70.23 (391.63) | 80.16 (643.85) | 77.7 (661.43) | 115.83 (1790.72)
  CD8-CD40L, Day 21 [N=111,41,109,34] | 3.9 (52.29) | 3.45 (30.93) | 5.61 (34.07) | 4.86 (162.75)
  CD8-IL-2, Day 21 [N=111,41,109,34] | 45.48 (251.49) | 57.71 (422.85) | 45.97 (342.71) | 77.59 (1217.04)
  CD8-INF-g, Day 21 [N=111,41,109,34] | 61.44 (390.6) | 62.56 (629.74) | 55.07 (661.84) | 95.39 (1777.86)
  CD8-TNF-a, Day 21 [N=111,41,109,34] | 55.42 (306.06) | 75.79 (579.85) | 63.94 (609.54) | 82.29 (1468.85)
  CD8 All doubles, Day 42 [N=120,43,118,29] | 77.73 (499.25) | 63.45 (462.64) | 79.56 (765.47) | 141.31 (2816.12)
  CD8-CD40L, Day 42 [N=120,43,118,29] | 5.32 (100.78) | 3.51 (24.09) | 5.23 (51.86) | 3.41 (253.17)
  CD8-IL-2, Day 42 [N=120,43,118,29] | 42.77 (261.13) | 40.01 (296.52) | 50.37 (413.85) | 97.06 (1832.58)
  CD8-INF-g, Day 42 [N=120,43,118,29] | 55.71 (506.29) | 64.19 (434.7) | 63.71 (767.88) | 119.73 (2845.99)
  CD8-TNF-a, Day 42 [N=120,43,118,29] | 59.51 (434.37) | 40.62 (375.13) | 59.1 (689.32) | 72.24 (2394.5)

35. Secondary Outcome: Geometric Mean of Influenza-specific Cluster of Differentiation (CD) 4/CD8 T-cells
Description: as for outcome 31
Time Frame: At Day 180
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: Cells
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 132 | 47 | 122 | 41
Cells
  CD4 All doubles [N=132,47,122,41] | 1247.34 (1000.47) | 760.03 (637.84) | 1515.07 (1982.71) | 850.48 (764.04)
  CD4-CD40L [N=132,47,122,41] | 1188.86 (939.31) | 729.72 (583.83) | 1455.68 (1789.27) | 808.25 (678.83)
  CD4-IL-2 [N=132,47,122,41] | 1172.16 (957.55) | 704.32 (596.04) | 1433.08 (1921.82) | 774.93 (742.9)
  CD4-INF-g [N=132,47,122,41] | 654.11 (661.08) | 461.8 (494.66) | 763.06 (1243.6) | 558.99 (654.35)
  CD4-TNF-a [N=132,47,122,41] | 937.82 (839.91) | 585.7 (578.22) | 1143.69 (1444.11) | 636 (713.19)
  CD8 All doubles [N=132,47,121,41] | 32.11 (293.81) | 23.66 (370.71) | 41.28 (753.94) | 36.77 (685.05)
  CD8-CD40L [N=132,47,121,41] | 2.04 (26.32) | 1.93 (31.43) | 2.47 (499.31) | 1.8 (23.59)
  CD8-IL-2 [N=132,47,121,41] | 18.78 (178.46) | 18.86 (269.95) | 23.7 (704.78) | 18.95 (465.37)
  CD8-INF-g [N=132,47,121,41] | 26.37 (288.43) | 28.27 (365.36) | 41.21 (663.4) | 28.29 (688.23)
  CD8-TNF-a [N=132,47,121,41] | 22.3 (270.88) | 20.94 (289.74) | 36.68 (390.84) | 40.55 (588.74)

36. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], headache, myalgia, shivering and sweating. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day follow-up period (Days 0 to 6) after any vaccination
Population: as for outcome 26
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
Number analyzed (Participants) | 164 | 61 | 159 | 51
Subjects
  Arthralgia | 13 | 5 | 13 | 1
  Grade 3 Arthralgia | 1 | 0 | 2 | 0
  Related Arthralgia | 0 | 1 | 2 | 0
  Fatigue | 32 | 7 | 39 | 6
  Grade 3 Fatigue | 2 | 2 | 6 | 0
  Related Fatigue | 1 | 1 | 8 | 0
  Fever (Axillary) >38.0°C | 2 | 1 | 5 | 0
  Fever (Axillary) ≥39.0°C | 1 | 1 | 1 | 0
  Related Fever | 0 | 1 | 1 | 0
  Headache | 27 | 6 | 34 | 2
  Grade 3 Headache | 0 | 1 | 1 | 0
  Related Headache | 2 | 3 | 6 | 0
  Myalgia | 24 | 5 | 28 | 3
  Grade 3 Myalgia | 1 | 0 | 4 | 1
  Related Myalgia | 2 | 1 | 4 | 0
  Shivering | 2 | 3 | 9 | 2
  Grade 3 Shivering | 1 | 0 | 1 | 0
  Related Shivering | 0 | 2 | 2 | 0
  Sweating | 16 | 8 | 19 | 2
  Grade 3 Sweating | 0 | 0 | 1 | 0
  Related Sweating | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs were collected within 21/30 days after the first/second vaccination. Solicited AEs were collected within 7 days after each vaccination. SAEs were collected for the entire study period (Day 0-Mth 24) within 4 timeframes: Days 0-51, Day 52-Month 6, Months 6-12 and Months 12-24. No unsolicited AEs with a frequency of >5% were reported (the number of participants at risk in the Other AE section is therefore the number of participants at risk analysed for the solicited AEs reporting)
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Arm/Group | GSK1562902A 1 Group | GSK1562902A 2 Group | GSK1562902A 3 Group | GSK1562902A 4 Group
All-Cause Mortality (participants affected / at risk) | 0/165 | 2/61 | 3/159 | 0/52
Serious Adverse Events (participants affected / at risk) | 19/165 | 11/61 | 16/159 | 5/52
Other Adverse Events (participants affected / at risk) | 69/164 | 8/61 | 75/159 | 6/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK1562902A 1 Group (N=165) | GSK1562902A 2 Group (N=61) | GSK1562902A 3 Group (N=159) | GSK1562902A 4 Group (N=52)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and 51 post vaccination.
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 — SAE reported between Day 0 and 51 post vaccination.
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 — SAE reported between Day 0 and 51 post vaccination.
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and 51 post vaccination.
Cardiac failure congestive (Cardiac disorders) | 0/164 | 1/58 | 1/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/164 | 0/58 | 0/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Atrial fibrillation (Cardiac disorders) | 1/164 | 0/58 | 0/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Cardiac failure acute (Cardiac disorders) | 0/164 | 0/58 | 1/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Cerebral hemorrhage (Vascular disorders) | 0/164 | 0/58 | 1/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Cerebral ischaemia (Nervous system disorders) | 1/164 | 0/58 | 0/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Cerebrovascular accident (Nervous system disorders) | 0/164 | 0/58 | 1/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Femoral neck fracture (Injury, poisoning and procedural complications) | 0/164 | 0/58 | 1/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/164 | 0/58 | 0/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Sciatica (Nervous system disorders) | 1/164 | 0/58 | 0/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Transient ischaemic attack (Nervous system disorders) | 0/164 | 1/58 | 0/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Ventricular fibrillation (Cardiac disorders) | 0/164 | 1/58 | 0/158 | 0/51 — SAE reported between Day 52 and 180 post vaccination.
Pneumonia (Infections and infestations) | 1/130 | 0/48 | 1/125 | 0/42 — SAE reported between Day 181 and Month 12 post vaccination.
Lobar pneumonia (Infections and infestations) | 0/130 | 0/48 | 0/125 | 1/42 — SAE reported between Day 181 and Month 12 post vaccination.
Lower limb fracture (Injury, poisoning and procedural complications) | 1/130 | 0/48 | 0/125 | 0/42 — SAE reported between Day 181 and Month 12 post vaccination.
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/130 | 0/48 | 0/125 | 0/42 — SAE reported between Day 181 and Month 12 post vaccination.
Phlebitis (Vascular disorders) | 0/130 | 0/48 | 1/125 | 0/42 — SAE reported between Day 181 and Month 12 post vaccination.
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/130 | 0/48 | 0/125 | 1/42 — SAE reported between Day 181 and Month 12 post vaccination.
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/130 | 0/48 | 1/125 | 0/42 — SAE reported between Day 181 and Month 12 post vaccination.
Schizophrenia (Psychiatric disorders) | 0/130 | 0/48 | 1/125 | 0/42 — SAE reported between Day 181 and Month 12 post vaccination.
Aortic aneurysm (Vascular disorders) | 0/122 | 1/45 | 1/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Acute myocardial infarction (Cardiac disorders) | 1/122 | 0/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Angioedema (Skin and subcutaneous tissue disorders) | 1/122 | 0/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Aortic valve incompetence (Cardiac disorders) | 0/122 | 1/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Arterial insufficiency (Vascular disorders) | 0/122 | 1/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/122 | 0/45 | 1/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Biliary colic (Hepatobiliary disorders) | 0/122 | 0/45 | 1/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Bradycardia (Cardiac disorders) | 1/122 | 0/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/122 | 1/45 | 0/117 | 0/36
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1/122 | 0/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Cholelithiasis (Hepatobiliary disorders) | 0/122 | 1/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Extrasystoles (Cardiac disorders) | 1/122 | 0/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Hip fracture (Injury, poisoning and procedural complications) | 0/122 | 0/45 | 0/117 | 1/36 — SAE reported between Month 12 and Month 24 post vaccination.
Inguinal hernia (Gastrointestinal disorders) | 0/122 | 1/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Intentional overdose (Injury, poisoning and procedural complications) | 0/122 | 1/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Intestinal obstruction (Gastrointestinal disorders) | 0/122 | 0/45 | 0/117 | 1/36 — SAE reported between Month 12 and Month 24 post vaccination.
Polyneuropathy (Nervous system disorders) | 1/122 | 0/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/122 | 0/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/122 | 0/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/122 | 0/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Renal failure (Renal and urinary disorders) | 0/122 | 0/45 | 1/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Venous insufficiency (Vascular disorders) | 0/122 | 0/45 | 1/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Cerebrovascular accident (Nervous system disorders) | 2/130 | 0/48 | 0/125 | 0/42 — SAE reported between Day 181 and Month 12 post vaccination.
Pneumonia (Infections and infestations) | 1/122 | 1/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24 post vaccination.
Cardiac failure acute (Cardiac disorders) | 0/122 | 1/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24.
Cardiac failure congestive (Cardiac disorders) | 0/122 | 0/45 | 1/117 | 0/36 — SAE reported between Month 12 and Month 24.
Cerebrovascular accident (Nervous system disorders) | 0/122 | 0/45 | 1/117 | 0/36 — SAE reported between Month 12 and Month 24.
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/122 | 0/45 | 0/117 | 0/36 — SAE reported between Month 12 and Month 24.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1562902A 1 Group (N=164) | GSK1562902A 2 Group (N=61) | GSK1562902A 3 Group (N=159) | GSK1562902A 4 Group (N=51)
Pain (General disorders) | 69 | 6 | 75 | 3
Induration (General disorders) | 10 | 0 | 15 | 0
Redness (General disorders) | 19 | 0 | 30 | 1
Swelling (General disorders) | 19 | 0 | 15 | 0
Arthralgia (General disorders) | 13 | 5 | 13 | 1
Fatigue (General disorders) | 32 | 7 | 39 | 6
Headache (General disorders) | 27 | 6 | 34 | 2
Myalgia (General disorders) | 24 | 5 | 28 | 3
Shivering (General disorders) | 2 | 3 | 9 | 2
Sweating (General disorders) | 16 | 8 | 19 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.